CLINICAL TRIAL: NCT06783283
Title: Transcranial Alternating Current Stimulation to Engage Theta-Gamma Coupling and Enhance Working Memory in Patients With Mild Cognitive Impairment
Brief Title: TACS to Engage Theta-Gamma Coupling and Enhance Working Memory in Patients With MCI (tACS-MCI)
Acronym: tACS-MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Soterix Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 056-2023
Record Dates: First submitted 2024-12-12; First posted 2025-01-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Memory Impairment; Executive Function; Transcranial Alternating Stimulation; Neuroplasticity; Electroencephalography; Working Memory; Cognition; Prefrontal Cortex; Transcranial Electrical Stimulation; Dementia; Alzheimer's Disease; Temporal Cortex
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: In a 1x1 factorial Randomized Controlled Trial (RCT), the investigators will randomize 20 MCI participants to one of the two treatment arms: tACS and sham-tACS, with 10 participants in each group. tACS will be delivered bilaterally to the PFC and temporal cortices. Each participant will receive daily stimulation for 10 days. Working memory and TGC during working memory performance will be assessed at baseline and following the last day of the study intervention. Working memory will be assessed using the N-back task and TGC using EEG during N-back performance.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be completed under triple-blind conditions. First, participants will be blind to whether they are randomized to the active treatment (tACS) or sham group (sham-tACS), which is achievable because it is difficult to distinguish the active treatment interventions from the control conditions. Second, the investigator team (investigators and interventionists delivering the 10-session course) will be blind to group assignment. Third, the outcomes assessors conducting the clinical, cognitive and EEG assessments at baseline and follow-ups will be blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tACS (Active Comparator): After completing the Baseline testing at Visit 1 and N-back EEG at Visit 2, MCI participants randomized to the active condition will receive a 10-session course of tACS (Visits 4-13), followed by a follow-up assessment, post intervention, at Visit 14.
  Interventions: Device: Transcranial Alternating Current Stimulation
- Sham tACS (Sham Comparator): After completing the Baseline testing at Visit 1 and N-back EEG at Visit 2, MCI participants randomized to the sham condition will receive a 10-session course of sham-tACS (Visits 4-13), followed by a follow-up assessment, post intervention, at Visit 14.
  Interventions: Device: Sham tACS

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Transcranial Alternating Current Stimulation (tACS) is a non-invasive electrical stimulation that will be used to stimulate the dorsolateral prefrontal cortex (dlPFC) and temporal cortices and in turn enhance Theta-Gamma Coupling (TGC) and working memory in Mild Cognitive Impairment (MCI). Each participant will receive daily stimulation for 10 days. To deliver the tACS, multiple electrodes embedded in a cap placed on the participant's head. Sham-tACS will follow the same procedure.
  Other Names: tACS
  Arms: Active tACS
Device: Sham tACS — During sham-tACS, the device will ramp up to the desired intensity over 60 seconds, and then will immediately ramp down, and the stimulation will be shut off, until the end of the session. At the end of the session, the device will again ramp up for 60 seconds and then ramp down. Sham-tACS will also target dlPFC and temporal cortices (similar to active). Each participant will receive daily sham-tACS for 10 days. To deliver the sham-tACS, multiple electrodes will be embedded in a cap placed on the participant's head.
  Arms: Sham tACS

SUMMARY:
This study is looking at a new non-invasive brain stimulation methods called transcranial alternating current stimulation (tACS) to see if it can improve working memory and thinking processes in people with Mild Cognitive Impairment (MCI). tACS is a low-risk, non-painful, low electrical current that circulates through the brain of awake participants and stimulates their brain cells. Participants must be 60 years of age and have a diagnosis of mild cognitive impairment. Participants will undergo treatment sessions that range from 1 to 1.5 hours at CAMH, 5 days a week, over a total of 2 weeks. In addition, participants will complete clinical and cognitive assessments and bloodwork at baseline and again after treatment.

DETAILED DESCRIPTION:
Current treatments for Alzheimer's disease dementia (AD) have limited efficacy probably because by the time AD is manifest it is too late to intervene. Thus, discovering interventions that will prevent AD is highly needed.

Mild Cognitive Impairment (MCI) is a condition that is considered a pre-stage to AD. In MCI, the frontal part of the brain supports the ability to compensate for memory problems which could delay progression to AD. This compensation is supported by "flexible" thinking which includes the ability to hold and manipulate information in mind for brief periods of time (e.g. doing mental math), also called working memory. Working memory has been shown by us and others to depend on the linking of brain waves across multiple brain waves frequencies.

Transcranial Alternating Current Stimulation (tACS) is a non-invasive electrical stimulation, applied to the scalp, that has been shown to improve this linking of brain waves in healthy older individuals. It has also been shown to enhance working memory in older individuals when this linking is enhanced. The effect of tACS on working memory and linking of brain waves in patients with MCI has not been demonstrated yet.

The study investigators propose to study the feasibility and preliminary effects of tACS on TGC and working memory in MCI participants. This proof-of-concept study will test whether tACS engages TGC as a target and, in turn, enhances working memory. Additionally, the investigators will explore the relationship among tACS effects and stress neuroreactivity and neuroimmune/inflammatory response (i.e., the interaction between the nervous system and the immune system), as well as the potential links with working memory.

If successful, our project will serve as a model for a larger trial to confirm the ability of tACS to prevent AD over multiple years of follow-up.

Objective 1: To determine the feasibility of tACS in older individuals with MCI. The investigators will examine recruitment and retention. Hypothesis 1a: At least 30% of screened participants will agree and be eligible to receive the intervention they are assigned to, i.e., tACS. Hypothesis 1b: At least 70% of participants will attend at least 80% of their treatment sessions.

Objective 2: To determine TGC engagement in response to tACS. The investigators will assess whether TGC increases in response to tACS. Hypothesis 2: Participants randomized to tACS will experience higher increase in TGC than those randomized to sham-tACS.

Objective 3: To determine change in working memory in response to tACS, and whether changes in TGC mediate changes in N-back performance with 2-back d' being the primary N-back outcome measure. Hypothesis 3a: Participants randomized to tACS will experience more improvement on N-back from baseline following the intervention than those randomized to sham-tACS. Hypothesis 3b: Across all participants, change in TGC will mediate change in N-back performance.

Exploratory Objective 4: To explore the relationships among tACS effects and stress neuroreactivity and neuroimmune/inflammatory response, as well as the potential links with working memory. Exploratory Hypothesis 4a: Baseline measure of stress neuroreactivity (i.e., salivary α-amylase and cortisol levels) will moderate response to tACS vs. sham-tACS. Exploratory Hypothesis 4b: Baseline measure of neuroimmune/inflammatory response (i.e., s100B, NSE, and MBP / IL-1β, IL-6, CRP, and TNF-α) will moderate response to tACS vs. sham-tACS. Exploratory Hypothesis 4c: Participants randomized to tACS will experience better stress neuroreactivity (i.e., salivary α-amylase and cortisol levels) from baseline following the intervention than those randomized to sham-tACS. Exploratory Hypothesis 4d: Participants randomized to tACS will experience better neuroimmune/inflammatory response (i.e., s100B, NSE, and MBP / IL-1β, IL-6, CRP, and TNF-α) from baseline following the intervention than those randomized to sham-tACS.

Exploratory Mediation Hypothesis: Across all participants, changes in stress neuroreactivity (i.e., salivary α-amylase and cortisol levels) and neuroimmune/inflammatory response (i.e., s100B, NSE, and MBP /I L-1β, IL-6, CRP, and TNF-α) will mediate change in TGC, N-back performance, and working memory.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or above,
2. Diagnosis of MCI due to AD using the core clinical criteria by the National Institute on Aging and Alzheimer's Association for MCI participants (NIA-AA) and ascertained by a study investigator. The following checklist will be used to ascertain the MCI diagnosis:

   1. Cognitive concern reflecting a change in cognition reported by patient or informant or clinician (i.e., historical or observed evidence of decline over time)
   2. Not demented ascertained using the study investigator opinion.
   3. No vascular, traumatic, or medical causes of cognitive decline ascertained using the study investigator opinion.
   4. Evidence of longitudinal decline in cognition, when feasible, and ascertained using the study investigator opinion.
3. Objective evidence of single or multi domain MCI, where single domain MCI refers to deficits using neuropsychology (NP) battery on only one of the cognitive domains (Speed of Processing; Working Memory; Executive Functioning; Verbal Memory; Visual Memory; Language) and multi domain MCI refers to deficits in more than one of these domains. To determine impairment in one or more cognitive domain, after the NP battery is administered and double scored, a consensus meeting will be held with the Research Analyst/Fellow, the study Principal Investigator and the study Neuropsychologist during which eligibility will be discussed. The meeting attendees will take into consideration the participant's education, parental education, pre-morbid IQ, physician's assessment and NP scores to determine if the participant has impairment in one or more cognitive domain.
4. Willingness to provide informed consent,
5. Ability to read and communicate in English (with corrected vision and hearing, if needed)

Exclusion Criteria:

1. Current use of an acetylcholine esterase inhibitor or memantine ascertained via participant's report, Medication List, or Electronic Medical Record (EMR).
2. Major Depressive Disorder with active symptoms in the last 3 months ascertained using the Mini International Neuropsychiatric Interview (MINI), or Structured Clinical Interview for DSM-5 (SCID), or EMR.
3. A lifetime diagnosis of bipolar disorder; intellectual disability; or a psychotic disorder ascertained using the MINI or SCID, or EMR.
4. Substance use disorder active in the last 3 months ascertained using the MINI or SCID, or EMR.
5. Any other DSM-5 diagnosis ascertained using the MINI or SCID, or EMR, that may be associated with prefrontal cortical dysfunction as ascertained using a study investigator opinion.
6. Current anticonvulsant use due to its impact on brain stimulation induced activity and ascertained using a Medication List or EMR. An exception will be made if they are taking gabapentin or pregabalin AND if the dose had been stable for at least 4 weeks prior to study entry AND if prescribed for chronic pain.
7. Current benzodiazepine use of more than what is equivalent to lorazepam 2 mg/day as ascertained using a Medication List. This is due to their known pro-GABAergic activity and the suppressive effect of GABAergic agents on cortical plasticity
8. Any contraindication to MRI or contraindication to tACS (e.g., cardiac pacemaker, acoustic device, history of seizures) ascertained using the tACS Safety Screen (tSS)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of All Screened Participants | Through treatment completion, at the end of 2-week intervention.
  Recruitment (percentage of all screened participants) will be examined.
  Hypothesis: At least 30% of screened participants will agree and be eligible to receive the intervention they are assigned to, i.e., tACS.
Percentage of All Enrolled Participants | Through treatment completion, at the end of 2-week intervention.
  Retention will be examined. Hypothesis: At least 70% of participants will attend at least 80% of their treatment sessions.

SECONDARY OUTCOMES:
Theta-gamma Coupling | Through treatment completion, at the end of 2-week intervention.
  The modulation index obtained from the EEG recording during N-Back
N-Back | Through treatment completion, at the end of 2-week intervention.
  Cognitive test via EEG measured by d', a sensitivity index based on the z scores of the hit and false alarm rates using the following formula: d' = z(H)- z(FA) where H is the hit rate and FA is the false alarm rate.
Mediation of TGC on changes in N-back performance | Through treatment completion, at the end of 2-week intervention.
  The beta value generated by Linear Model examining the association between changes in TGC and changes in N-back performance.

OTHER OUTCOMES:
PASAT | Through treatment completion, at the end of 2-week intervention.
  Modified Paced Auditory Serial Addition Test (PASAT) test total correct responses across both types of trials
Neuroimmune response | Through treatment completion, at the end of 2-week intervention.
  Measured by concentration of s100B, NSE (pg/mL) in blood sample
Neuroimmune response | Through treatment completion, at the end of 2-week intervention.
  Measured by concentration of MBP (ng/mL) in blood sample.
Inflammatory response | Through treatment completion, at the end of 2-week intervention.
  Measured by concentration of IL-1β, IL-6, CRP, and TNF-α (pg/mL) in salivary sample.
Stress neuroreactivity | Through treatment completion, at the end of 2-week intervention.
  Measured by the dynamics of α-amylase and cortisol levels across baseline phase (before PASAT) and response phase (after PASAT); the intercept, baseline slope, and response slope

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kumar, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication can be shared upon a reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publishing the results of the study.
Access Criteria: New proposals approved by ethics board, data will be shared using Centre for Addiction and Mental Health databank.

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research